CLINICAL TRIAL: NCT02838927
Title: Epi-Hypo: Survey on Epidemiology of Hypoparathyroidism in France
Brief Title: Survey on Epidemiology of Hypoparathyroidism in France
Acronym: Epi-Hypo
Status: Recruiting | Type: Observational
Sponsor: European Georges Pompidou Hospital (Other)
Collaborators: Oscar - Filière Santé Maladies Rares (Unknown)
Responsible Party: Principal Investigator, Jean-philippe Bertocchio, MD, PhD, MD, PhD, European Georges Pompidou Hospital
Other Study IDs: EpiHypo
Record Dates: First submitted 2016-07-09; First posted 2016-07-20 (Estimated); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Hypoparathyroidism
Keywords: Hypoparathyroidism; Epidemiology; Medication Therapy Management
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypoparathyroidism: No intervention.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Very few data has been published on the epidemiology of hypoparathyroidism worldwide: none exists specifically for France. Hypoparathyroidism could led to complications. Here, the investigators plan to collect data about both epidemiology, medication and complication of hypoparathyroidism in France.

DETAILED DESCRIPTION:
Very few data has been published on the epidemiology of hypoparathyroidism worldwide. None exists specifically in France. Hypoparathyroidism could led to complications: e.g. symptomatic hypocalcemia, calcifications (brain, eye and other soft tissues), nephrolithiasis/nephrocalcinosis, renal insufficiency. Here,the investigators plan to collect data about both epidemiology, medication and complication of hypoparathyroidism in France.

ELIGIBILITY:
Inclusion Criteria:

* patient fro whom chronic hypoparathyroidism is diagnosed
* patient living in France

Exclusion Criteria:

* patient who does not want his data to be collected in this registry
* pseudo-hypoparathyroidism
* acute hypoparathyroidism

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients for whom hypoparathyroidism is diagnosed in France
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of the epidemiology of patients with hypoparathyroidism in France | Through study completion, about 2 years
  Data collected by questionnaire about etiology of hypoparathyroidism, filled by physicians from clinic folders

SECONDARY OUTCOMES:
Assessment of the biology at inclusion will describe the evolution of the included population from diagnosis to now (inclusion) | At inclusion (under treatment): through study completion, about 2 years
  Number of patients with at least one anomaly at biology (calcemia in mM, calciuria in mmol/j, parathormone in pg/ml, creatininemia in µM, phosphatemia in mM, vitamin D in nmol/l & magnesemia in mM) at inclusion
Assessment of the management at inclusion will describe treatment and complications at inclusion | At inclusion (under treatment): through study completion, about 2 years
  Number of patients with clinical outcomes (complications such as cataract, nephrolithiasis, nephrocalcinosis, and others) and their management at inclusion
Assessment of the biology (calcemia, calciuria, parathormone, creatininemia, phosphatemia & magnesemia) at diagnosis and drug therapy at inclusion will describe population | Through study completion, about 2 years
  Number of patients with at least one anomaly at biology (calcemia in mM, calciuria in mmol/j, parathormone in pg/ml, creatininemia in µM, phosphatemia in mM, vitamin D in nmol/l & magnesemia in mM) at diagnosis

OTHER OUTCOMES:
Assessment of the physician's management will help describing the habits of french physician who manage hypoparathyroidism in terms of follow-up | At inclusion
  Data on habits of included physicians about their management of patients with hypoparathyroidism: frequency of complications' follow-up (nephrocalcinosis, cataract, nephrolithiasis and other calcifications) in terms of radiology (CT-scan, echotomography, radiography) and biology (calcium in mM, phosphate in mM, parathormone in pg/ml, magnesium in mM, vitamin D in nmol/l and creatininemia in µM).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Bertocchio, MD, PhD, Principal Investigator — European Georges Pompidou Hospital, APHP
Locations (57):
- France (57):
  - Felix Guyon Hospital, Saint-Denis, La Réunion
  - Hôpital Privé de Provence, Aix-en-Provence
  - Amiens University Hospital, Amiens
  - Clinic Auch Area, Auch
  - Henri Mondor Hospital, Aurillac
  - Jean Minjoz Hospital, Besançon
  - Blanquefort, Blanquefort
  - Avicenne Hospital, AP-HP, Bobigny
  - Jean Verdier Hospital, AP-HP, Bondy
  - University Hospital, Bordeaux
  - Bourgoin Jallieu Hospital, Bourgoin
  - La Cavale Blanche Hospital, Brest
  - Côte de Nacre Hospital, Caen
  - Henri Mondor Hospital, APHP, Créteil
  - Dax-Côte d'Argent Hospital, Dax
  - University Hospital, Dijon
  - Grenoble Alpes Hospital, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - Kremlin-Bicêtre Hospital, APHP, Le Kremlin-Bicêtre
  - Le Mans Hospital, Le Mans
  - Libourne Hospital, Libourne
  - Claude Huriez Hospital, Lille
  - Edouard Herriot Hospital, HCL, Lyon
  - La Conception Hospital, AP-HM, Marseille
  - Clinic Metz Area, Metz
  - Mercy Hospital, Metz
  - Clinic area, Mérignac
  - Arnaud de Villeneuve Hospital, Montpellier
  - Brabois Hospital, Nancy
  - University Hospital, Nantes
  - University Hospital, Nice
  - Georges Renon Hospital, Niort
  - Caremeau Hospital, Nîmes
  - European Georges Pompidou Hospital, APHP, Paris
  - Clinic Paris Area, Paris
  - Cochin Hospital, APHP, Paris
  - Lariboisière Hospital, APHP, Paris
  - Necker Hospital, AP-HP, Paris
  - Pitié-Salpêtrière Hospital, APHP, Paris
  - Saint-Louis Hospital, AP-HP, Paris
  - Tenon Hospital, APHP, Paris
  - Passy Hospital, Passy
  - Clinic Poitiers Area, Poitiers
  - Laennec Hospital, Quimper
  - Reims University Hospital, Reims
  - Clinic Rennes Area, Rennes
  - Charles Nicolle Hospital, Rouen
  - Saint Florent Le Vieil, Saint-Florent-le-Vieil
  - Clinic Area, Saint-Junien
  - Clinique du Landy, Saint-Ouen
  - Hautepierre Hospital, Strasbourg
  - Sainte Anne Hospital, HIA, Toulon
  - Larrey Hospital, Toulouse
  - Guy Chatiliez Hospital, Tourcoing
  - Bretonneau Hospital, Tours
  - Valenciennes Hospital, Valenciennes
  - CHIV - Lucie et Raymond Aubrac, Villeneuve-Saint-Georges

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bertocchio JP, Grosset N, Groussin L, Kamenicky P, Larceneux F, Lienhardt-Roussie A, Linglart A, Maruani G, Mirallie E, Pattou F, Seervai RNH, Sido C, Silve C, Vilfaillot A, Tabarin A, Vantyghem MC, Houillier P. Practice patterns for chronic hypoparathyroidism: data from patients and physicians in France. Endocr Connect. 2022 Jan 31;11(1):e210350. doi: 10.1530/EC-21-0350. PMID 34939939